CLINICAL TRIAL: NCT03427593
Title: Phenotype-genotype Correlation in a Sub-population of Severe Primary Immunodeficiency With Lymphoproliferation and Neutropenia
Brief Title: Severe PID With Lymphoproliferation and Neutropenia
Acronym: DICEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6642
Record Dates: First submitted 2018-01-15; First posted 2018-02-09 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Primary Immune-Deficiency (PID) Common Variable Immune Deficiency (CVID)
Keywords: CVID; Neutropenia; Autoimmunity; Lymphoproliferation
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Common Variable Immunodeficiency; Neutropenia; Autoimmune Diseases | interventions — High-Throughput Nucleotide Sequencing; Exome Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients (Experimental): Patients with the phenotype (PID and Neutropenia and lymphoproliferation)
  Interventions: Genetic: FACS analyses; Genetic: Target Sequencing by NGS ( Next-generation sequencing); Genetic: Whole Exome Sequencing
- relatives (parents) (Other)
  Interventions: Genetic: FACS analyses; Genetic: Target Sequencing by NGS ( Next-generation sequencing); Genetic: Whole Exome Sequencing
- Controls (Sham Comparator)
  Interventions: Genetic: FACS analyses

INTERVENTIONS:
Genetic: FACS analyses — FACS analyses
Genetic: Target Sequencing by NGS ( Next-generation sequencing) — Target Sequencing by NGS ( Next-generation sequencing)
  Arms: Patients; relatives (parents)
Genetic: Whole Exome Sequencing — Whole Exome Sequencing
  Arms: Patients; relatives (parents)

SUMMARY:
The purpose of this study is to analyse the phenotype in a sub-population of adults with severe primary immunodeficiency with lymphoproliferation and neutropenia and to decipher the possible pathways involved, especially under the hypothesis of a CTLA4/LRBA schema

ELIGIBILITY:
Inclusion Criteria :

* >18 years old
* CVID (Common Variable Immunodeficiency)
* Neutropenia
* Lymphoproliferation

Exclusion Criteria :

- Secondary immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Identification of known mutations by target sequencing of all known genes involved in CVID phenotypes. | Day 0 (inclusion)
  Target-NGS
Identification of new mutations in new genes in CVID by WES (whole exome sequencing) strategy. | Day 0 (inclusion)
  WES (Whole exome sequencing), If no known mutations is founded by T-NGS
Validation or not of a pathological pathway involving CTLA4/LRBA or a related pathway in T-cells. Validation by the mean of functional analysis of T-cells in vitro of CTLA4 expression and response to stimulation. RNA-sequencing in sorted cells. | Day 0 (inclusion)

SECONDARY OUTCOMES:
Deciphering of new possible genes involved in the phenotype : Patient without known mutation in genes involved in PID will benefit of an extended analyse of the WES to find a possible condidate genes | Day 0 (inclusion)
  After WES analyses

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Immunologie Clinique et VIH - Hôpital Civil, Strasbourg, France

REFERENCES:
- [Result] Guffroy A, Mourot-Cottet R, Gerard L, Gies V, Lagresle C, Pouliet A, Nitschke P, Hanein S, Bienvenu B, Chanet V, Donadieu J, Gardembas M, Karmochkine M, Nove-Josserand R, Martin T, Poindron V, Soulas-Sprauel P, Rieux-Laucat F, Fieschi C, Oksenhendler E, Andre-Schmutz I, Korganow AS; DEFI study group. Neutropenia in Patients with Common Variable Immunodeficiency: a Rare Event Associated with Severe Outcome. J Clin Immunol. 2017 Oct;37(7):715-726. doi: 10.1007/s10875-017-0434-2. Epub 2017 Aug 26. PMID 28842786